CLINICAL TRIAL: NCT00862420
Title: A Randomized, Double Blind, Parallel Group Study to Investigate the Safety of 12 Weeks of Clopidogrel 75 mg/Day Versus Ticlopidine 200 mg/Day in Patients With Peripheral Arterial Disease - With Extended Treatment of Clopidogrel 75 mg/Day for 40 Weeks
Brief Title: Safety Evaluation of Clopidogrel Sulfate in Patients With Peripheral Arterial Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SFY10810
Record Dates: First submitted 2009-03-09; First posted 2009-03-16 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Peripheral Arterial Disease (PAD)
Keywords: Platelet aggregation inhibitors; Peripheral arterial disease (PAD)
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Clopidogrel; Ticlopidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clopidogrel (Experimental): 75 mg clopidogrel once daily from Day 1 to Week 12
  Interventions: Drug: clopidogrel (SR25990)
- Ticlopidine (Active Comparator): 200 mg ticlopidine once daily from Day 1 to Week 12
  Interventions: Drug: ticlopidine

INTERVENTIONS:
Drug: clopidogrel (SR25990) — oral administration (tablets)
  Arms: Clopidogrel
Drug: ticlopidine — oral administration (tablets)
  Arms: Ticlopidine

SUMMARY:
Primary objective:

* To evaluate whether 12 weeks of clopidogrel is superior to ticlopidine in terms of lower risk of the safety events of interests in patients with peripheral arterial disease (PAD)

Secondary objectives:

* To compare the risk of bleeding adverse events, serious adverse events and overall safety of clopidogrel with ticlopidine
* To compare the risk of vascular events of clopidogrel with ticlopidine
* To document the long-term safety of clopidogrel for a total of 52 weeks
* To document the vascular events of clopidogrel for a total of 52 weeks

ELIGIBILITY:
Inclusion Criteria:

Documented symptomatic peripheral arterial disease (one or both of the following two primary criteria must be satisfied):

* Current intermittent claudication with Ankle Brachial Index (ABI) < 0.90
* A history of intermittent claudication together with previous related intervention in a leg

Exclusion Criteria:

* Patients who had acute atherothrombotic events or any invasive therapies within 30 days before the randomization, or patients who planned any invasive therapies within 12 weeks after the randomization
* Bleeding diathesis, coagulopathy and present bleeding disease
* Previous intracranial bleeding or hemorrhagic stroke
* Uncontrolled hypertension

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2009-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Safety events of interest including clinical significant bleeding, blood disorders, hepatic dysfunction and other serious adverse drug reactions (death, hospitalization...) | Week 12 (on treatment)

SECONDARY OUTCOMES:
Bleeding adverse events, Serious adverse events, Overall safety | Week 12, 52 (on treatment)
Vascular events | Week 12, 52 (on study)
Safety events of interest (see above) | Week 52 (on treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Shigematsu, Head Professor/MD/PhD, Principal Investigator — Second Department of Surgery (Vascular Surgery), Tokyo Medical University
Locations (1):
- Sanofi-Aventis Administrative Office, Tokyo, Japan

REFERENCES:
- [Derived] Shigematsu H, Komori K, Tanemoto K, Harada Y, Nakamura M. Clopidogrel for Atherothrombotic Event Management in Patients with Peripheral Arterial Disease (COOPER) Study: Safety and Efficacy of Clopidogrel versus Ticlopidine in Japanese Patients. Ann Vasc Dis. 2012;5(3):364-75. doi: 10.3400/avd.oa.12.00039. PMID 23555538